CLINICAL TRIAL: NCT02432898
Title: Non-Invasive Imaging of the Human Eye
Status: Withdrawn | Type: Observational
Why Stopped: No subjects were enrolled in this protocol
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: Topcon-001-2014
Record Dates: First submitted 2014-11-20; First posted 2015-05-04 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Willing and Able Subjects for Ocular Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal Healthy Eyes: Normal healthy eyes with no known ocular diseases
  Interventions: Device: 3D OCT-1; Device: 3D OCT-2000; Device: DRI OCT-1; Device: NW-300; Device: CT-1P; Device: TRK-2P; Device: SP-1P; Device: SL-D701; Device: MC-4S

INTERVENTIONS:
Device: 3D OCT-1 — Spectral Domain OCT Device
Device: 3D OCT-2000 — Spectral Domain OCT Device
Device: DRI OCT-1 — Swept Source OCT Device
Device: NW-300 — Fundus Camera
Device: CT-1P — Tonometry
Device: TRK-2P — Tonometry, Corneal Topography
Device: SP-1P — Specular Microscopy
Device: SL-D701 — Slit Lamp Imaging
Device: MC-4S — Visual Acuity Testing

SUMMARY:
Evaluate the clinical information obtained from the use of the machines.

DETAILED DESCRIPTION:
Evaluate the clinical information provided by these devices and determine their clinical utility and efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients from 18 to 80 years old who have full legal capacity to volunteer on the date the informed consent is signed.
2. Subjects who can follow the instructions by the clinical staff at the clinical site and can attend examinations on the scheduled examination date.

Exclusion Criteria:

1. History of ocular pathology.
2. History of cataract of ocular surgical procedures that render the cornea opaque or otherwise impact its ability to be imaged using the investigational device.
3. History of systemic disease
4. fixation problems which may prevent obtaining good quality images in the eye.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal subjects will be recruited from Topcon Medical Systems.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Device Evaluation | 1 Hour
  Determine Clinical Utility, Efficacy, and Safety

CONTACTS AND LOCATIONS:
Overall Officials: Danny Leung, Principal Investigator — Topcon Corporation
Locations (1):
- Topcon Medical Systems, Inc., Oakland, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided